CLINICAL TRIAL: NCT00046501
Title: Morning LANTUS v. Intermediate-acting Insulin 2x/Day as Basal Insulin in a Multiple Daily Inj. w/ Humalog in Adolescents w/ Type 1 Diabetes Mellitus: an Active-controlled, Open, Randomized, Gender-stratified, Two-arm, Parallel-group Study
Brief Title: Compare Blood Sugar Level Between Lantus in the Morning and Other Insulins in Type 1 Diabetes Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4030
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Injections; Isophane Insulin, Human; insulin, long-acting, human; Insulin Lispro

INTERVENTIONS:
Drug: Lantus (insulin glargine [rDNA origin] injection)
Drug: Humulin N
Drug: Humulin L
Drug: Lispro

SUMMARY:
The purpose of the study is to compare the effect in blood sugar control between Lantus and twice daily intermediate acting insulins (NPH or Lente) when used as the basal insulin in a multiple daily injection setting with fast acting insulin (Lispro)

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes treated with insulin only for at least 1 year,
* with a Tanner stage of ≥ 2,
* had evidence of decreased insulin secretory capacity (fasting C-peptide concentration ≤0.5 mmol/L) and 7.0%≤A1c≤9.5% at screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250
Dates: Start 2002-11; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
to measure change in glycemic control as measured by hemoglobin A1c (A1c). | from baseline to endpoint (last available post-treatment assessment)

SECONDARY OUTCOMES:
Change in A1c | from baseline to individual study time points
Percentage of subjects achieving an A1c ≤7.0; percent of preteens (12 years and below) achieving 8%; teens (13-18 years) achieving 7.5% | During the study conduct
Change in fasting self-monitored blood glucose (SMBG) for weekdays, weekends and weekday/weekend combined | from baseline to endpoint
Change in urinary spot random microalbumin-to-creatinine (A/C) ratio | from baseline to endpoint
Change in 8-point blood glucose profiles for weekdays, weekends, and weekday/weekend combined | from baseline to endpoint
Change in average basal insulin doses | from baseline to endpoint
Change in lipids (total cholesterol [TC], high-density lipoprotein cholesterol [HDL], low-density lipoprotein cholesterol [LDL], and triglycerides [TGs]) | from baseline to endpoint
Change in glucose | from baseline to endpoint
Occurrence of hypoglycemia | from the informed consent signature to the end of the study
Adverse events (AEs) | from the informed consent signature to the end of the study
Clinical values: physical examination, vital signs, change in age-adjusted body mass index (BMI) | from the informed consent signature to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Doug Green, Study Director — Sanofi
Locations (1):
- Aventis, Bridgewater, New Jersey, United States